CLINICAL TRIAL: NCT06199206
Title: The Effect of Therapeutic Play on Children's Anxiety and Fear Levels and Parents' Anxiety Levels Before Lumbar Puncture Procedure in Children Aged 6 - 12 Years
Brief Title: The Effect of Therapeutic Play on Children's Anxiety and Fear Before Lumbar Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assist. Prof., Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-46059653-050.99-232013695
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Anxiety and Fear
Keywords: theraputic play; lumbar punction; children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Before the procedures, therapeutic games will be played with the children and people of the intervention groups with eLPi dolls and other play materials prepared in accordance with anatomy. The parent will be with the child during this game, which will be played in his/her own room.
  Interventions: Other: Theraputic Play
- Control Group (No Intervention): No therapeutic play will be made to children. Children will be verbally informed about the lumbar puncture.

INTERVENTIONS:
Other: Theraputic Play — Before the procedures, therapeutic games will be played with the children and people of the intervention groups with eLPi dolls and other play materials prepared in accordance with anatomy. The parent will be with the child during this game, which will be played in his/her own room.
  Arms: Intervention Group

SUMMARY:
The study will be conducted with the randomized controlled experimental method. The children who attended the pediatric department will divide into two groups via randomization in the computer environment. After random selection, children in the intervention group will play a therapeutic game before the lumbar puncture procedure. Children in the control group will not undergo any procedure before the lumbar puncture procedure. Parents will be present with their children in both groups during the procedure. While the child's anxiety and fear level is measured, the parent's anxiety level will also be measured.

DETAILED DESCRIPTION:
For the child, illness and hospitalization are frightening, disturbing and unpleasant situations. Children are more fragile and sensitive than adults because they are inadequate to meet their health care needs and have not completed sufficient physical, cognitive and social development. Whether the disease is acute or chronic, the pain or limitation of movement it causes, the need for isolation, the child's previous hospitalization and stress experiences, the state of preparation for hospitalization, the anxiety level of family members and intra-family relationships affect the child's response to the disease and hospitalization. Medical interventions performed in a hospital environment are among the stimuli that create psychological and physiological stress in the child. It has been determined that children are not given effective education before medical procedures, and children who do not receive adequate preparation experience increased fear and anxiety, and experience problems such as feelings of insecurity and rejection of interventions. In addition, this experience causes the child to develop negative reactions to later hospital experiences. One of the medical interventions performed on children in the hospital environment is lumbar puncture (LP). Lumbar puncture is a method that has been used by different disciplines for diagnosis and treatment purposes for years. When the LP procedure is performed on children compared to adults, it may cause more anxiety and fear in both the child and their parents. Increased levels of anxiety and fear may cause children and parents to reject the procedure. Nurses have important roles in reducing the stress, anxiety and fear of children and their parents during these medical procedures. In line with the family-centered care philosophy, nurses should inform the child and their parents about the procedure and prepare the child for the procedure with methods such as therapeutic games. With the therapeutic play method, the child's negative emotions such as fear and anxiety regarding the procedure can be managed. This research will be conducted to determine the effect of therapeutic play applied to children between the ages of 6 and 12, who are admitted to the pediatric ward, before the LP procedure, on the children's anxiety and fear levels and their parents' anxiety levels.

The sample size of the study has been determined by the power analysis (G*Power 3.1), in line with the results obtained from the studies which have been conducted using a similar research method. The sample size was found to be a total of 28 children including minimum of 14 children for each group. It was estimated that case losses may occur and therefore, it was decided to conduct the study with a total of 34 children including 17 children in two groups. Children who meet the average selection criteria prior to data collection will be identified. Verbal and written permission will be obtained from the children of the selected students to participate, and verbal consent will be obtained from the children through the 'Informed Voluntary Consent Form'.

LP storage in children in both control and intervention periods; Routine practices in the clinic will be carried out before, during and after the procedure. Written consent will be given for the procedure. For those who do not agree to have the LP procedure, intermittent oral feeding (solid oral intake for two hours, liquid oral intake for six hours) will be discontinued and preparations for the procedure will be made.

No application will be made to reveal the fear and anxiety levels of the control groups. Only children and their parents will be informed about the transaction. Five minutes before the procedure within the scope of the research, the "State-Trait Anxiety Inventory" and "Children's Fear Scale" for children and the "Beck Anxiety Scale" for parents will be evaluated. Intervention Group: Children in the intervention group and their parents will play therapeutic games with specially prepared eLPi dolls and other play materials before the procedure. The parent will be with the child during this game, which will be played in the child's own room and bed. Before the procedure, the "State-Trait Anxiety Inventory" and the "Children's Fear Scale" will be used for children and the "Beck Anxiety Scale" will be used for parents. Therapeutic play steps; First, the child's temperature will be measured with a thermometer on one of the eLPi dolls of his/her own choosing. An oxygen mask will be attached to the doll with a high fever, it will be positioned, and some liquid will be drawn into the syringe from balls containing liquid placed on the back in accordance with the anatomy. After covering the back area with gauze, that liquid will be examined with the child under the toy microscope. After the therapeutic game, the child will enter the sterilely prepared intervention room with the child. Before the LP procedure, the activity of the child's vascular access will be checked, an oxygen mask will be applied and monitored. During the LP procedure, the child will be positioned and sedation planned according to the child's weight will be administered intravenously. After the CSF samples are taken, the blood sugar level will be checked. The area where the LP procedure is performed will be covered with gauze for twenty-four hours. After the LP procedure, the patient will be kept in the intervention room for thirty to forty-five minutes to ensure that the sedation wears off and the child's general condition is observed. One hour after the LP procedure, the anxiety of children in both the intervention and control groups will be determined with the "State-Trait Anxiety Inventory" scale, and the children's fear will be determined with the "Children's Fear Scale". Additionally, the "Beck Anxiety Scale" will be applied to determine the anxiety level of the parents.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 and 12,
* Children do not have any work, speech, mental or mathematical problems,
* Before LP was performed, children,
* Inclusion of parents and children who do not agree to participate voluntarily.

Exclusion Criteria:

* Children under 6 years old and over 12 years old,
* Children with hearing, speech, mental or neurological problems,
* Children who have had LP before,
* Parents and their children who do not agree to participate in the research will be excluded from the research.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Children's Anxiety Level (State-Trait Anxiety Inventory for Children-CDSSI) | 45 minutes before lumbar punction, 10 minutes before lumbar punction and 1 hour after lumbar punction
  Developed by Spielberger (1976), this performance has two optional subscales for state and trait anxiety, each consisting of 20 questions. Points are given as 0, 1 or 2 depending on the protection of the substance. Situational anxiety; It consumes the individual's free anxiety, covering specific circumstances at a decisive time, and may vary according to external factors. Trait anxiety reflects the individual's general absence and the individual's anxieties in general. Cronbach's Alpha was 0.82, reflecting state anxiety. In the study; If trait anxiety will not be used, the section on state anxiety appropriate to the learning method will be used. 20 questions are asked and there are 3 options for each question. Questions will earn between one and three points. The highest score that can be obtained from the scale is 60 and the lowest score is 20. The scale score is reached at the point where state anxiety occurs.
Children's Fear Level (Children's Fear Scale-CFS) | 45 minutes before lumbar punction, 10 minutes before lumbar punction and 1 hour after lumbar punction
  It is used to measure the child's fear level. The one-item scale consists of 5 facial expressions, regardless of gender. It is a scale that evaluates between 0 and 4, consisting of showing five drawn facial expressions ranging from neutral expression (0 = no anxiety) to scared face (4 = severe anxiety). It was created based on the Faces Anxiety Scale, developed by Mc Kinley et al. (2003) to measure the fear or anxiety of adults in the intensive care unit. Cronbach's alpha value was reported to be 0.89.

SECONDARY OUTCOMES:
Mother's Anxiety Level (Beck Anxiety Scale) | 45 minutes before lumbar punction, 10 minutes before lumbar punction and 1 hour after lumbar punction
  It is a Likert-type self-rating scale, developed by Aaron Beck (1988), consisting of 21 items and used to determine the frequency of anxiety symptoms experienced by individuals, with each item scored between "0 - 3". Cronbach's alpha value was reported to be 0.94. When the total score on the scale is between "0 - 7" points, anxiety is minimal, "8 - 15" points is mild, "16 - 25" points is moderate, and "26 - 63" points is severe. It is considered as anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Erkut, PhD, Principal Investigator — Maltepe University
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No